CLINICAL TRIAL: NCT05732597
Title: How to Decide Which COVID-19 Patient With Myocardial Infarction to Send to the Cath Lab? - A Case Series of COVID-19 Patients With Myocardial Infarction
Brief Title: Acute Coronary Syndrome in Patients With COVID-19
Acronym: ACS-COVID
Status: Completed | Type: Observational
Sponsor: Bulgarian Cardiac Institute (Network)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2023-02-16; First posted 2023-02-17 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Myocardial Infarction; Acute Coronary Syndrome; COVID-19; Myocardium; Injury
Keywords: COVID-19; Coronavirus; Acute coronary syndrome; Troponin
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; COVID-19; Wounds and Injuries; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with ACS and no IRA: Patients with acute coronary syndrome (ACS) during a COVID-19 infection, who after undergoing coronary angiography - no infarct-related artery (IRA) is found
  Interventions: Procedure: Coronary angiography
- Patients with ACS and IRA: Patients with acute coronary syndrome (ACS) during a COVID-19 infection, who after undergoing coronary angiography - an infarct-related artery (IRA) is found
  Interventions: Procedure: Coronary angiography

INTERVENTIONS:
Procedure: Coronary angiography — A coronary angiogram is a procedure that uses X-ray imaging to see the patient's blood vessels of the heart. The test is generally done to see if there's a restriction in blood flow going to the heart.

SUMMARY:
The aim of this study was to find a clinical or laboratory parameter, that would help in distinguishing between COVID-19 patients with myocardial infarction (MI), who have an infarct-related artery (IRA) and therefore, require immediate revascularization, and those, who have no IRA.

DETAILED DESCRIPTION:
The coronavirus pandemic has hit the world with its vast contagiousness, high morbidity, and mortality Apart from the direct damage to the lung tissue, the corona virus infection is associated with multiple organ damage, including the heart. Emerging evidence reveals a direct correlation between COVID-19 and cardiovascular complications, such as heart failure, myocarditis, arrhythmias, conduction abnormalities and acute coronary syndromes. The SARS-CoV-2 infection can frequently induce coagulation abnormalities that are associated with cardiopulmonary deterioration and death as a possible complication in all patients, despite presence or absence of concomitant risk factors and diseases. In addition, many patients with severe COVID-19 undergo thromboembolic events, which seem to be related to this particular coagulopathy. One of the most unpleasant and life-threatening types of thromboembolism is the one involving the coronary circulation, thus causing a heart attack. Many additional problems arise due to this condition e.g., access to a Cath lab, exposure of additional medical personnel, more complications and increased mortality for the patients.

Invasive angiography for COVID-19 patients is logistically challenging and, in some cases, there is no intervention target, since microcirculatory disease and thrombosis is common in this group. Therefore, the investigators studied in detail the case series of 10 patients referred for primary percutaneous coronary intervention (pPCI) for MI in our catheterization laboratory during the course of COVID-19 infection. And the investigators set themselves the purpose to evaluate if there are some factors or parameters that could predict the presence of an interventional target - infarct related artery (IRA), prior to catheterization, and to determine their sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Acute coronary syndrome (ACS)
* COVID-19 infection

Exclusion Criteria:

* No combination of ACS and COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient above 18 years old with ACS and COVID-19 infection
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-02-27 (Actual); Study Completion 2022-02-27 (Actual)

PRIMARY OUTCOMES:
to find a clinical or laboratory parameter, that would help in distinguishing between COVID-19 patients with MI and IRA and those, who have no IRA | During the whole study

CONTACTS AND LOCATIONS:
Locations (1):
- Heart and brain center of clinical excellence, University hospita, Pleven, Bulgaria, Pleven, Bulgaria

IPD SHARING:
Plan to Share IPD: No